CLINICAL TRIAL: NCT02888314
Title: Pokemon Go and Physical Activity Online Survey
Brief Title: Pokemon Go and Physical Activity
Acronym: Pokemon
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00075789
Record Dates: First submitted 2016-08-06; First posted 2016-09-05 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-09

CONDITIONS: Physical Activity
Keywords: mHealth; Pokemon Go
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study to evaluate the association between Pokemon Go and physical activity through a survey among Pokemon Go players.

DETAILED DESCRIPTION:
Pokemon Go is a location-based reality mobile game for iOS and Android devices developed by Niantic. Making use of GPS and the camera of compatible devices, the game allows players to capture virtual creatures, called Pokemon, who appear on cellphone screens as though in the real world. In order to search and capture the Pokemon, the players needs to go out and become more active. For this reason, the game has great potential to promote physical activity. Nevertheless, there has no study evaluating the potential impact of Pokemon Go on physical activity. The investigator proposes a retrospective online survey. Participants are instructed to enter data of their daily physical activity as reported in iPhone Health App. Number of "Steps" and % greater than 10,000 steps/day will be compared before and after installing the Pokemon Go app.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who use iPhone and have played Pokemon Go before July 31, 2016 and agree to consent to participate in the survey

Exclusion Criteria:

* Subjects who do not use iPhone
* Have not played Pokemon Go before July 31, 2016
* Unable to provide informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who use iPhone and have played Pokemon Go before July 31, 2016
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2016-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Average number of steps per day | Between June 15 and July 31, 2016
  Number of steps as reported on the iPhone Health app
Change in number of steps after Pokemon Go | From June 15 to July 31, 2016, assessed up to 6 weeks
  Differences in number of steps per day before and after Pokemon Go

SECONDARY OUTCOMES:
Greater than 10,000 steps per day | Between June 15 and July 31, 2016
  Percent of days in which subjects reached greater than 10,000 steps/day

CONTACTS AND LOCATIONS:
Overall Officials: Ying Ying, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xian Y, Xu H, Xu H, Liang L, Hernandez AF, Wang TY, Peterson ED. An Initial Evaluation of the Impact of Pokemon GO on Physical Activity. J Am Heart Assoc. 2017 May 16;6(5):e005341. doi: 10.1161/JAHA.116.005341. PMID 28512111